CLINICAL TRIAL: NCT04179617
Title: Impact of New Product Standards for JUUL Among Dual JUUL/Combusted Cigarette Users
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Enrollment was never initiated; COVID prevented participant enrollment
Sponsor: Duke University (Other)
Collaborators: University of Michigan (Other); Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Pro00103010
Record Dates: First submitted 2019-11-08; First posted 2019-11-27 (Actual); Last update posted 2021-08-25 (Actual); Status verified 2020-09

CONDITIONS: Smoking; E-cigarette Use; Cigarette Smoking
Keywords: JUUL; dual use; multiple tobacco product use; nicotine content; tobacco regulatory science
MeSH Terms: conditions — Smoking; Vaping; Cigarette Smoking

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Preferred nicotine content JUUL pod (Experimental): During one experimental visit, participants will have access to a JUUL loaded with a 5% nicotine content pod (their preferred pod)
  Interventions: Other: 5% nicotine content JUUL pod
- Low nicotine content JUUL pod (Experimental): During one experimental visit, participants will have access to a JUUL loaded with a 3% nicotine content pod (non-preferred pod)
  Interventions: Other: 3% nicotine content JUUL pod

INTERVENTIONS:
Other: 5% nicotine content JUUL pod — JUUL pods that contain 5% nicotine
  Arms: Preferred nicotine content JUUL pod
Other: 3% nicotine content JUUL pod — JUUL pods that contain 3% nicotine
  Arms: Low nicotine content JUUL pod

SUMMARY:
To date the majority of experimental tobacco regulatory science has focused specifically on the impact of possible tobacco product standards (e.g. limiting e-cigarette flavor) on the use of the single tobacco product targeted by the standard (e.g. e-cigarettes) among individuals who primarily or solely use the targeted product (e.g. vapers). Whereas this "single target" approach has yielded a large amount of actionable evidence, it has also resulted in a significant gap in the regulatory science evidence base for two reasons: First, the focus on single tobacco product users has resulted in very little evidence regarding the impact of possible new product standards among multiple tobacco product (MTP) users. MTP users make up a sizeable proportion (30-40%) of the tobacco using population and individuals who use e-cigarettes (EC) and combusted cigarettes (CC) comprise the largest MTP using group (40% of MTP users). A lack of data on this population means that estimates of the impact of new product standards on public health are incomplete.

Despite some data derived from hypothetical tasks, little experimental research exists to evaluate how potential tobacco regulations might impact the use of other tobacco products in addition to the targeted product. It is critical to anticipate how potential restrictions on the EC market may impact EC and other tobacco product-such as CC-use.

In the proposed research, we will recruit young adult (age 21-29) dual EC/CC users evaluate the demand for participants' usual brand CC as compared to EC that vary in nicotine content (e.g., 5% vs. 3% pods). Participants will engage in a validated concurrent choice task in which they will work for fixed doses of EC vapor or CC smoke in exchange for expended effort. In addition, we will seek to answer this question in samples of dual EC and CC users-individuals who, because they regularly use both EC and CC, are most vulnerable to changes in the appeal of EC and CC brought about by a product standard limiting EC flavors.

DETAILED DESCRIPTION:
The Food and Drug Administration (FDA) can enact tobacco product standards. Under the Family Smoking Prevention and Tobacco Control Act (FSPTCA), the FDA Secretary has the authority to "adopt tobacco product standards… if the Secretary finds that a tobacco product standard is appropriate for the protection of the public health" based on evidence of the "risks and benefits to the population as a whole…". To date, substantial tobacco regulatory science (TRS) research has been conducted to inform new standards, including research on the impact of the nicotine content in CC and e-cigarettes (EC) products.

Significant gaps exist in the extant TRS knowledge base. Despite the large amount of actionable evidence generated to date, most TRS has taken a "single target" approach. Research has focused on the impact of possible tobacco product standards (e.g., nicotine reduction in CC) on the use of the single tobacco product targeted by the standard (i.e., CC) among individuals who primarily or solely use the targeted product (i.e., CC smokers). This approach has resulted in significant gaps in the TRS evidence base in two important ways: First, the focus on single tobacco product users has resulted in little evidence regarding the impact of new product standards on multiple tobacco product (MTP) users. MTP constitute 30-40% of the tobacco using population; dual EC and CC users comprise 44% of MTP users (Preliminary Studies). As such, dual EC/CC users represent a substantial minority of tobacco product users. A lack of data on this population means that estimates of the potential impact of new product standards on public health are incomplete.

Second, regulations targeting one product will likely impact other tobacco products, as well. In our recent work, we present evidence that any two tobacco products vary in the degree to which they substitute for one another and hypothesize that new standards targeting one product may have "off-target" effects impacting the appeal and use of other products. This is the central premise of this research. We hypothesize that the degree of substitution between two products varies, at least in part, as a function largely of product characteristics (e.g. flavor, nicotine strength). For instance, prior research (and Preliminary Studies) indicate that the availability of flavored e-liquid may determine the degree to which EC serve as a substitute for CC among both current and former CC users, suggesting that a limit on e-liquid flavors would reduce EC substitutability for CC.

Finally, the size of the dual EC/CC using population and degree of substitutability between EC and CC products have important implications for determining the population health impact of new standards for tobacco products. There is general agreement that EC and CC exist along a continuum of risk with combusted products (including CC) exposing the user to greater amounts of toxicants relative to non-combusted products (including EC). Thus, it is possible that two individuals, both of them dual EC/CC users, have similar levels of nicotine dependence and nicotine exposure, but very different toxicant exposure due to differences in the relative amounts of EC and CC used. Putatively then, new product standards that alter the appeal and use of either EC or CC can similarly increase or decrease toxicant exposure by changing the amount of each product used.

We propose that changes in one product (e.g., EC) can result in changes in the appeal and use of another product (e.g., CC), thus altering the degree to which one substitutes for another-a research question that has received comparatively little attention, but is critical for informing FDA regulation. We will systematically and experimentally evaluate the: a) the smoking and vaping topography and appeal of participants' usual brand (UB) CC and JUUL EC that vary in nicotine content (Aim 1); b) effects of limiting EC nicotine content on preferences for users' usual brand of CC (Aim 2); and c) potential moderators of product preferences (Aim 3).

JUUL brand EC are of particular interest for a number of reasons. JUUL-a pod-based EC-entered the U.S. market in 2015, and has skyrocketed in popularity. As of 2018, JUUL had 72% of the U.S. EC market share-a 453% increase over 2016. JUUL provides similar nicotine delivery to CC and can be used discreetly. Finally, these low wattage systems are typically used with e-liquids containing nicotine salts, which allow for e-liquid with higher nicotine concentrations to be consumed with less harshness than freebase nicotine. The increasing popularity of JUUL EC, along with their potential for significant nicotine delivery, highlights the need for research concerning this product. We also propose to conduct this research among a sample of dual JUUL EC and CC users-individuals who, because they regularly use both JUUL EC and CC, are most vulnerable to changes in the appeal of JUUL EC and CC brought about by a product standard limiting EC nicotine content.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 21-29 inclusive;
* Combusted cigarette smoker for ≥3 months AND smoke combusted cigarettes ≥1 day/past week;
* Owner and user of JUUL brand e-cigarette for ≥3 months AND use JUUL ≥1 day/ past week;
* Current or previous use of JUUL branded pods;
* Breath alcohol level=0.000;
* Provided contact information for 2 individuals who can corroborate JUUL EC and CC use
* Willing to abstain from EC and CC use for 24 hours prior to Experimental Visits

Exclusion Criteria:

* Reporting that 3% nicotine content JUUL pods are their preferred nicotine content;
* Reporting that nicotine-free pods are their preferred pod;
* Vaping THC or CBD concentrates (e.g., oils, waxes, shatters, crumbles) in the past 3 months;
* Pregnant, trying to become pregnant, breastfeeding;
* Plans to quit using e-cigarettes or regular cigarettes in the next 30 days;
* Current use of smoking cessation aids or participation in smoking cessation treatment;
* Allergies to propylene glycol or glycerin;
* Lung or breathing problems (e.g., asthma, COPD, bronchitis) within the past 3 months;
* Systolic blood pressure ≥160 mmHg;
* Diastolic blood pressure ≥100 mmHg;
* Heart rate ≥115 bpm

Ages: 21 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2021-10 (Estimated); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Participant rating of how much they liked the product | Within 2 minutes of sampling product(s)
  Participants are asked the question: "How much do you like the product?" and asked to rate it on a scale from 0-100 (0 = not at all, 100 = extremely)
Participant rating of whether or not they would use the product again | Within 2 minutes of sampling product(s)
  Participants are asked the question: "Would you use it again?" and asked to rate it on a scale from 0-100 (0 = not at all, 100 = definitely)
Participant rating of how much they would pay for a day's worth of the product | Within 2 minutes of sampling product(s)
  Participants are asked the question: "How much would you pay for a day's worth?" and asked to rate it on a scale from $0-$100
Mean puff volume taken when using JUUL | Measurements taken over the course of a 5-minute window during the Appeal Phase
  A topography device will measure the volume of the 4 puffs taken when using JUUL during the Appeal Phase of the study; an average of the volume of these 4 puffs will be calculated
Mean puff volume taken when using combusted cigarettes | Measurements taken over the course of a 5-minute window during the Appeal Phase
  A topography device will measure the volume of the 4 puffs taken when using a combusted cigarette during the Appeal Phase of the study; an average of the volume of these 4 puffs will be calculated
Number of ratios completed for JUUL | The number of ratios completed will be calculated over a 1-hour period during the Reinforcement Phase
  The number of ratios completed (during a Progressive Ratio Task) to earn a puff of JUUL will be calculated
Number of ratios completed for combusted cigarettes | The number of ratios completed will be calculated over a 1-hour period during the Reinforcement Phase
  The number of ratios completed (during a Progressive Ratio Task) to earn a puff of a combusted cigarette will be calculated

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Pacek, PhD, Principal Investigator — Duke University

IPD SHARING:
Plan to Share IPD: No